CLINICAL TRIAL: NCT00002767
Title: PHASE III TRIAL OF MELACINE PLUS INTERFERON ALFA-2B VERSUS INTERFERON ALFA-2B IN PATIENTS WITH DISSEMINATED MALIGNANT MELANOMA
Brief Title: Interferon Alfa With or Without Vaccine Therapy in Treating Patients With Metastatic Melanoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: GlaxoSmithKline (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000064732; CORIXA-2885-14; RIR-2885-14; YALE-HIC-8666; NCI-V96-0883
Record Dates: First submitted 1999-11-01; First posted 2004-09-02 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2007-05

CONDITIONS: Melanoma (Skin)
Keywords: stage IV melanoma; recurrent melanoma
MeSH Terms: conditions — Melanoma | interventions — detox adjuvant; Interferon-alpha

INTERVENTIONS:
Biological: Detox-B adjuvant
Biological: recombinant interferon alfa

SUMMARY:
RATIONALE: Interferon alfa may interfere with the growth of cancer cells.Vaccines may make the body build an immune response to kill tumor cells. It is not yet known whether melanoma vaccine plus interferon alfa is more effective than interferon alfa alone in treating patients with metastatic melanoma.

PURPOSE: Randomized phase III trial to compare the effectiveness of interferon alfa with or without vaccine therapy in treating patients with metastatic melanoma.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare survival following immunotherapy with an allogeneic melanoma vaccine plus interferon alfa-2b (IFN-A) vs. IFN-A alone in patients with metastatic melanoma. II. Assess the safety and toxicity of immunotherapy with an allogeneic melanoma vaccine plus IFN-A in these patients. III. Compare the frequencies of durable complete responses in each treatment group. IV. Compare overall clinical objective response, duration of response, and time to disease progression in each treatment group. V. Compare the effects of immunotherapy with an allogeneic melanoma vaccine plus IFN-A vs IFN-A alone on quality of life in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are stratified by location of metastatic sites (visceral and bone vs nonvisceral and lung) and number of metastatic sites (1 vs 2 vs 3 or more). Patients are randomized to one of two treatment arms. Arm I: Patients receive allogenic melanoma cell lysate vaccine with detoxified endotoxin subcutaneously (SQ) weekly on weeks 1-5 and 8-12. Interferon alfa (IFN-A) SQ is administered three times a week beginning on week 4. Patients with responding or stable disease receive vaccine monthly beginning on week 16. IFN-A continues in the absence of disease progression or unacceptable toxicity. Arm II: Patients receive IFN-A SQ three times a week beginning on week 1. Treatment continues in the absence of disease progression or unacceptable toxicity. Quality of life is assessed before, during, and after treatment. Patients are followed every 3 months.

PROJECTED ACCRUAL: Approximately 300 patients will be entered over 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed malignant melanoma that is metastatic (any pT, any N, M1 by AJCC staging) Measurable disease by physical exam or noninvasive radiologic procedure No concurrent or prior diagnosis of ocular melanoma No CNS metastases No patients who can be rendered NED by surgery unless patient declines surgery

PATIENT CHARACTERISTICS: Age: 18 and over Performance status: ECOG 0 or 1 Life expectancy: At least 4 months Hematopoietic: Absolute granulocyte count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin no greater than 2 mg/dL AST or ALT no greater than 3 times normal No evidence of hepatic failure No active hepatitis Renal: Creatinine clearance at least 40 mL/min Cardiovascular: No myocardial infarction within 6 months No decompensating congestive heart failure No unstable angina No current symptomatic arrhythmia Other: No known HIV antibody No thyroid abnormality uncontrollable by medication No medical, sociological, or psychological impediment to study compliance No pre-existing psychiatric condition (especially depression) or history of severe psychiatric disorder No autoimmune disease (e.g., systemic lupus erythematosus, multiple sclerosis, ankylosing spondylitis) No concurrent malignancy except nonmelanomatous skin cancer Not pregnant or nursing Negative pregnancy test Effective contraception required of fertile women No history of egg allergies

PRIOR CONCURRENT THERAPY: Biologic therapy: At least 12 months since interferon alfa or melanoma vaccine No prior immunotherapy for metastatic disease No concurrent cytokines or levamisole Chemotherapy: No prior chemotherapy for metastatic disease At least 4 months since adjuvant therapy No concurrent chemotherapy Endocrine therapy: At least 1 week since corticosteroids No concurrent immunosuppressives (e.g., azathioprine or cyclosporine) Radiotherapy: Prior radiotherapy for metastatic disease allowed Surgery: See Disease Characteristics Prior surgery for metastatic disease allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 1996-01

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth B. Von Eschen, PhD, Study Chair — GlaxoSmithKline
Locations (27):
- United States (27):
  - University of Alabama Comprehensive Cancer Center, Birmingham, Alabama
  - Beckman Research Institute, City of Hope, Duarte, California
  - University of California San Diego Cancer Center - La Jolla, La Jolla, California
  - Kaiser Permanente Medical Center - Oakland, Oakland, California
  - Kaiser Permanente Medical Center-Sacramento, Sacramento, California
  - UCSF Cancer Center and Cancer Research Institute, San Francisco, California
  - Kaiser Permanente Medical Group - San Francisco, San Francisco, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente Medical Center - Vallejo, Vallejo, California
  - University of Connecticut Health Center, Farmington, Connecticut
  - Yale Comprehensive Cancer Center, New Haven, Connecticut
  - Sylvester Cancer Center, University of Miami, Miami, Florida
  - Adventist Health System/Sunbelt, Inc., Orlando, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Lutheran General Cancer Care Center, Park Ridge, Illinois
  - University of Louisville Hospital, Louisville, Kentucky
  - Creighton University Cancer Center, Omaha, Nebraska
  - Norris Cotton Cancer Center, Lebanon, New Hampshire
  - University of New Mexico Cancer Research & Treatment Center, Albuquerque, New Mexico
  - Interlakes Oncology/Hematology PC, Rochester, New York
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Barrett Cancer Center, The University Hospital, Cincinnati, Ohio
  - Christ Hospital, Cincinnati, Ohio
  - CCOP - Columbus, Columbus, Ohio
  - Hematology Oncology Consultants Inc, Columbus, Ohio
  - Oregon Cancer Center at Oregon Health Sciences University, Portland, Oregon
  - Southwest Regional Cancer Center, Austin, Texas